CLINICAL TRIAL: NCT06197737
Title: Effects of Moderate Intensity Interval Training and Sprint Interval Training on Patients Having Chronic Asthma.
Brief Title: Specific Modified Exercise Program for Patients Having Chronic Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/MS-PT/01379
Record Dates: First submitted 2023-05-04; First posted 2024-01-09 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — High-Intensity Interval Training; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate Intensity Interval Training (Experimental): These participants will perform moderate intensity interval training. The intervention will be applied thrice a week. Moderate intensity interval training in which they do stair climbing 3 times a week And for every 1 interval I will ask them to take rest for 3 minutes.
  Interventions: Other: Moderate Intensity Interval Training
- Sprint Interval Training (Experimental): These participants will perform sprint interval training and frequency will be 3 days a week.
  The participants will perform sprint interval training in which they will do stair climbing 3 times a week with a fast pace.
  Interventions: Other: Sprint Interval Training
- pharmacological treatment (Other): They will be on pharmacological treatment as prescribed by their pulmonologist.
  Interventions: Other: pharmacological treatment

INTERVENTIONS:
Other: Moderate Intensity Interval Training — Participants in this group will perform moderate intensity interval training in which they will perform stair climbing 3 times a week and for every 1 interval I will ask them to take rest for 3 minutes.
  Arms: Moderate Intensity Interval Training
Other: Sprint Interval Training — sprint interval training in which they will do stair climbing 3 times a week with a fast pace.
  Arms: Sprint Interval Training
Other: pharmacological treatment — They will be on pharmacological treatment as prescribed by their pulmonologist.
  Arms: pharmacological treatment

SUMMARY:
To compare the effects of moderate intensity interval training and sprint interval training on patients having chronic asthma.

DETAILED DESCRIPTION:
Chronic asthma is a complex heterogeneous disease characterized by multiple aggravating factors. Asthma is treated with two types of medicines , long term medicines and quick relieve medicine. Although the relationship between asthma and the effects of HIIT/SIT were studied in the literature, there was not one comparing the results of these aforementioned studies. The purpose of this study is to find the effects of moderate intensity interval training and sprint interval training on pat determine effects of group wise physical activity on asthma related quality of life. To determine the effects of group wise physical activity on cardiorespiratory endurance

ELIGIBILITY:
Inclusion Criteria:

* Patients having chronic asthma
* Age between 15-25 years.
* Participants having no dyspnea at rest .
* Participants scoring 13 or less on borg scale
* Exclusion Criteria
* History of co-morbidities.
* History of recent fractures.
* Participants scoring greater than 13 on BORG scale

Exclusion Criteria:

* Exercise induced asthma (evaluated through BRUCE protocol).
* Individuals with co-morbidities related to any neurological, cardiovascular, psychological and musculoskeletal disorders .
* Patients score falling 15 or more on Borg scale.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Assessment of change in the Inspiratory Capacity | Baseline, 8th week and then 16th week
  It will measured using an incentive spirometer
Assessment of change in the Pulmonary Function | Baseline, 8th week and then 16th week
  Electronic spirometer will be used to measure all the parameters of pulmonary function.
Assessment of change in the Oxygen saturation | Baseline, 8th week and then 16th week
  Measured using pulse oximeter before, during and after the intervention.
Assessment of change in the Rate of perceived exertion / dyspnea | Baseline, 8th week and then 16th week
  measured through borg scale during the assigned intervention
Assessment of change in the cardiovascular endurance | Baseline, 8th week and then 16th week
  PACER test for cardiovascular endurance test

CONTACTS AND LOCATIONS:
Overall Officials: Malik Muhammad Ali Awan, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Abasyn University, Islamabad, Federal Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No